CLINICAL TRIAL: NCT07174895
Title: Efficacy of Tranexamic Acid With/Without Drain in Knee Arthroplasty: A Study From Northwest Syria
Brief Title: Tranexamic Acid and Drain Use in Knee Arthroplasty
Acronym: TNAKnee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Idlib University (Other)
Responsible Party: Principal Investigator, Mhmoud Adnan Al salamah, Principal Investigator, Department of Orthopedic Surgery, Idlib University, Idlib University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T.A in Knee Arthroplasty; NW-Syria-TKA-Study-01 (Other: Idlib University)
Record Dates: First submitted 2025-08-30; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Osteoarthritis, Knee
Keywords: Arthroplasty, Replacement, Knee Tranexamic Acid Blood Loss, Surgical Drainage Perioperative Care Hemostasis, Surgical Randomized Controlled Trial
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Tranexamic Acid; Suction

STUDY DESIGN:
Intervention Model Description: > This is a prospective randomized clinical trial including 192 patients undergoing total knee arthroplasty. Participants were randomly assigned to one of three groups to assess the effects of intra-articular tranexamic acid and/or suction drainage on total and hidden blood loss, transfusion requirements, postoperative limb swelling, wound-related complications, and knee range of motion.
Masking Description: Not applicable. The study was conducted as an open-label trial with no blinded parties.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tranexamic Acid with Suction Drainage (Experimental): Patients undergoing total knee arthroplasty received intra-articular injection of 3 g tranexamic acid diluted in 100 mL normal saline after wound closure. A closed suction drain was inserted intra-articularly and subcutaneously, activated two hours postoperatively.
  Interventions: Drug: Intra-articular Tranexamic Acid + Suction Drainage
- Tranexamic Acid without Drainage (Experimental): Patients undergoing total knee arthroplasty received intra-articular injection of 3 g tranexamic acid diluted in 100 mL normal saline after wound closure. No suction drain was used in this group.
  Interventions: Drug: Intra-articular Tranexamic Acid
- Suction Drainage without Tranexamic Acid (Active Comparator): Patients undergoing total knee arthroplasty had a closed suction drain inserted intra-articularly and subcutaneously, activated two hours postoperatively. No tranexamic acid was administered in this group.
  Interventions: Device: Suction Drainage Only

INTERVENTIONS:
Drug: Intra-articular Tranexamic Acid + Suction Drainage — Patients received intra-articular injection of 3 g tranexamic acid in 100 mL normal saline after wound closure, along with a closed suction drain inserted intra-articularly and subcutaneously, activated two hours postoperatively.
  Arms: Tranexamic Acid with Suction Drainage
Drug: Intra-articular Tranexamic Acid — Patients received intra-articular injection of 3 g tranexamic acid in 100 mL normal saline after wound closure. No suction drain was used.
  Arms: Tranexamic Acid without Drainage
Device: Suction Drainage Only — Patients had a closed suction drain inserted intra-articularly and subcutaneously, activated two hours postoperatively. No tranexamic acid was administered.
  Arms: Suction Drainage without Tranexamic Acid

SUMMARY:
This prospective randomized clinical study is designed to evaluate the effects of intra-articular tranexamic acid (TNA), with or without suction drainage, on perioperative blood management in patients undergoing total knee arthroplasty (TKA) for degenerative arthritis. A total of 192 patients will be randomly assigned to three groups: Group 1 will receive TNA with suction drainage, Group 2 will receive TNA only, and Group 3 will receive suction drainage only.

The primary outcomes will be total blood loss and transfusion requirements. Secondary outcomes will include hidden blood loss, drainage volume, postoperative limb swelling, wound-related complications, and knee range of motion. The study will help clarify whether suction drainage is necessary when intra-articular TNA is used during TKA.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is commonly associated with significant perioperative blood loss, which may increase transfusion requirements and associated risks such as immunologic reactions, infection, and delayed recovery. Tranexamic acid (TNA) is an antifibrinolytic agent that inhibits fibrinolysis by blocking the activation of plasminogen. Suction drainage is frequently used to prevent hematoma formation, but its benefit in reducing transfusion needs remains controversial.

This single-center, prospective randomized study will enroll 192 patients undergoing unilateral TKA for degenerative arthritis. Participants will be assigned to three groups: (1) TNA with suction drainage, (2) TNA only, and (3) suction drainage only. TNA will be administered intra-articularly at a dose of 3 g in 100 mL normal saline after wound closure. When applied, suction drains will be activated two hours postoperatively.

The primary outcomes will be total blood loss and transfusion requirement. The secondary outcomes will include hidden blood loss, drainage volume, postoperative limb swelling, wound-related complications, and knee range of motion at two months. Statistical analysis will be conducted using ANOVA, repeated-measures t-tests, and chi-square tests, with significance set at p ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients with degenerative knee arthritis
* Scheduled for unilateral total knee arthroplasty

Exclusion Criteria:

* Rheumatoid arthritis
* Cardiovascular diseases (e.g., angina, myocardial infarction, arrhythmia, cerebrovascular events)
* Coagulation disorders or thromboembolic disorders
* Severe infections
* Other serious health issues

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Total Blood Loss | Within 72 hours after surgery
  Total blood loss calculated using changes in hemoglobin concentration and the Good et al. formula.

SECONDARY OUTCOMES:
Hidden Blood Loss | Within 72 hours after surgery
  Hidden blood loss calculated as total blood loss minus drainage volume.
Drainage Volume | 24 hours postoperatively
  Total drainage collected through suction drains when applicable.
Number of Blood Transfusions | During hospital stay (up to 7 days postoperatively)
  Number of patients receiving blood transfusions based on NIH Consensus criteria (Hb < 8.0 g/dL, or <10.0 g/dL with symptoms).
Postoperative Limb Swelling | 1, 2, 4, and 6 weeks postoperatively
  Change in limb circumference at thigh, knee, and calf compared with preoperative baseline.
Wound-related Complications | Within 6 weeks after surgery
  Incidence of wound-related issues, including infection, hematoma, erythema, or superficial wound complications.
Thromboembolic Events (DVT/PE) | Within 6 weeks after surgery
  Incidence of deep vein thrombosis (DVT) confirmed with Doppler ultrasonography and pulmonary embolism (PE) if suspected clinically.
Postoperative Knee Range of Motion | 2 months postoperatively
  Range of motion measured with a goniometer (flexion and extension).

CONTACTS AND LOCATIONS:
Overall Officials: Mhmoud Adnan Al-Salamah, Principal Investigator — Idlib University
Locations (1):
- Faculity of Medicine, Idlib, Syria

REFERENCES:
- [Background] Hishimura R, Onodera T, Ohkoshi Y, Okada K, Matsuoka M, Matsubara S, Iwasaki K, Kondo E, Iwasaki N. The effect of local injection of tranexamic acid into peri-articular tissue versus drain clamping in total knee arthroplasty: a randomized controlled trial. BMC Musculoskelet Disord. 2022 Feb 2;23(1):111. doi: 10.1186/s12891-022-05058-6. PMID 35109837
- [Background] Kim MK, Ko SH, Nam YC, Jeon YS, Kwon DG, Ryu DJ. Optimal Release Timing of Drain Clamping to Reduce Postoperative Bleeding after Total Knee Arthroplasty with Intraarticular Injection of Tranexamic Acid. Medicina (Kaunas). 2022 Sep 5;58(9):1226. doi: 10.3390/medicina58091226. PMID 36143903
- [Background] Liu CH, Chang CH, Chang YH, Shih HN, Hu CC. Topical Fibrin Sealant (Tisseel@) Does Not Provide a Synergic Blood-Conservation Effect with Tranexamic Acid in Total Knee Arthroplasty-A Prospective Randomized Controlled Trial. Medicina (Kaunas). 2023 Nov 26;59(12):2078. doi: 10.3390/medicina59122078. PMID 38138181
- [Background] Zhang W, Li N, Chen S, Tan Y, Al-Aidaros M, Chen L. The effects of hypotensive anesthesia and regional anesthesia on intraoperative blood loss in total knee arthroplasty. World J Emerg Surg. 2024;19(1):33. doi:10.1186/s13017-024-00554-7
- [Background] Chaiyakit P, Kabkaew P, Hongku N, Wattanapreechanon P. Comparison of total blood loss between limited tourniquet use and conventional tourniquet use in total knee arthroplasty: a randomized controlled trial. BMC Musculoskelet Disord. 2024 Nov 15;25(1):918. doi: 10.1186/s12891-024-08058-w. PMID 39548417
- [Background] Zhou C, Gao X, Han H, Wang L, Jiang H. The efficacy and safety of tranexamic acid in primary total knee arthroplasty: a systematic review and meta-analysis. J Orthop Surg Res. 2024;19(1):37. doi:10.1177/15563316231208716.
- [Background] Liu Y, Ai J, Teng X, Huang Z, Wu H, Zhang Z, Wang W, Liu C, Zhang H. Risk factor analysis and establishment of a nomogram model to predict blood loss during total knee arthroplasty. BMC Musculoskelet Disord. 2024 Jun 10;25(1):459. doi: 10.1186/s12891-024-07570-3. PMID 38858713
- [Background] Gonzalez-Pola R, Tafoya-Olivos RO, Culebras-Almeida LA, Zermeño-Garcia G, Herrera-Lozano A. Minimizing bleeding and transfusion in single-stage bilateral hip and knee arthroplasty: a systematic review of current interventions. Rev Esp Cir Ortop Traumatol (Engl Ed). 2025;69(2):e58. doi:10.1016/j.recot.2025.02.002.
- [Background] Ju Y, Liu H, Jiang W, Huang Q, Zhou Z, Pei F. Perioperative blood loss of sequential administration of hemocoagulase Agkistrodon and Tranexamic acid for primary total knee arthroplasty: a randomized controlled trial. J Orthop Surg Res. 2025 May 13;20(1):457. doi: 10.1186/s13018-025-05867-0. PMID 40355919
- [Background] Liangliang L, Wei H, Tao Z, Pin P, Lianying H. Efficacy and safety of tranexamic acid in reducing hidden blood loss during unilateral total knee arthroplasty: a retrospective study. Front Med (Lausanne). 2025 Jun 3;12:1552893. doi: 10.3389/fmed.2025.1552893. eCollection 2025. PMID 40529153